CLINICAL TRIAL: NCT01476709
Title: Photonic Needle and Intraforaminal Epidural Injection (Sleeve) - Observational Study in Humans
Brief Title: Photonic Needle and Sleeve Study
Acronym: PhotonicNeedle
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: MEC 11-1-005
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Puncture; Instrument; Pain
Keywords: Puncture; Instrument; Optics and Photonics; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: evaluate the potential of the photonic needle (photonic needle technology) to discriminate tissues that are relevant to recognize during intraforaminal (transforaminal) epidural injection on lumbar level.

Objective: The primary objective of this study is to investigate the potential of the photonic needle to discriminate between correct and incorrect placement of the needle tip in the target area of the procedure (M4 - tissue), as confirmed by contrast-enhanced fluoroscopy. The secondary objectives are to investigate the differences in the optical signals obtained with the photonic needle at a set of different pre-defined positions (M1, M2 and M3) encountered along the needle trajectory during above-mentioned procedures, and to detect potential intravascular positioning of the needle-tip at the target point (M4 - blood), Study design: this is a single blind observational study. Study population: Patients who have radicular pain on lumbar level, for example caused by disc herniation, and/or lateral recessus stenosis and/or radiculopathy eci.

Main study parameters/endpoints: The main study parameters are: 1) successfully acquired diffuse reflectance spectra obtained at measurement point M4: midforaminal, halfway the foramen (the target treatment location) as encountered during image-guided intraforaminal injections on lumbar level, 2) confirmation of target area with fluoroscopy and injection of contrast fluid (gold standard), 3) "Certainty score" on a 3-point scale (1 = uncertain, 2 = certain, 3 = very certain) will be provided by the physician. The type of tissue present at the needle tip will be based on the information available from imaging .

The secondary study parameters are: 1) successfully acquired diffuse reflectance spectra obtained at measurement points M1-M3: M1 in muscle, M2 extra-foraminal, M3 foraminal at a distance 1/3 of the diameter of the foramen from the entrance of the foramen, as encountered during image-guided intraforaminal injections on lumbar level, 2) successfully acquired diffuse reflectance spectra obtained at measurement point M4, in case of a vascular puncture (M4-blood), 3) confirmation images by ultrasound imaging at location M1 as described above, 4) confirmation images by fluoroscopy at locations M2 and M3, 5) digital subtraction angiography images after contrast injection at location M4, confirming vascular penetration (gold standard for vessel puncture), 6) "Certainty score" on a 3-point scale (1 = uncertain, 2 = certain, 3 = very certain) provided by the physician for assignment of the type of tissue present at the needle tip, based on the information available from imaging at M1 and at M4.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for regular treatment: intraforaminal epidural injection
* Patients' age is 18 - 80 years
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Photodynamic therapy used before
* Inability to give informed consent
* Contrast fluid allergy
* Any operation on the spine at the side of intervention
* Coagulation disorders / disturbance
* Infections at the level of intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have radicular pain on lumbar level, caused by disc herniation, and/or lateral recessus stenosis and/or radiculopathy eci.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Statistical analysis of the difference between diffuse reflectance spectra obtained for correct and incorrect needle placement in the target area of the procedure. | direct measurement

SECONDARY OUTCOMES:
Statistical analysis of differences between diffuse reflectance spectra obtained in muscle, extra-foraminal, foraminal at a distance 1/3 of the diameter of the foramen from the entrance of the foramen,intravascular. | direct measurement

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van Kleef, prof. Dr., Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands